CLINICAL TRIAL: NCT04296513
Title: High-Definition White Light Endoscopy vs Optical Enhancement With High Definition Optical Magnification in the Diagnosis of Gastritis, H. Pylori Infection and Atrophic Gastritis in Dyspeptic Patients: A Randomized Controlled Trial.
Brief Title: Diagnosis of Gastritis, H. Pylori Infection and Atrophic Gastritis in Dyspeptic Patients
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED-02012020
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Gastritis, Atrophic; Helicobacter Pylori Infection; Intestinal Metaplasia; Gastritis
Keywords: endoscopy; gastritis
MeSH Terms: conditions — Gastritis, Atrophic; Gastritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gastric mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-Definition white light endoscopy.: evaluation of the gastric mucosa with high-definition white-light endoscopy (EG-29i10 gastroscope and EPKi7010 video processor). The endoscopy images will be seen on a 27inch, flat panel, high definition LCD monitor (Radiance™ ultraSC-WU27-G1520 model) by one endoscopist, randomly assigned via esophagogastroduodenoscopy.
  Interventions: Diagnostic Test: High-Definition white light endoscopy.
- High-definition magnification with digital chromoendoscopy.: The subject will be evaluated by upper endoscopy with the OE System (EPK-i7010 HD Video Processor and MagniView™ EG-2990Zi Video Gastroscope) with intravenous sedation in a standardized manner. This technique involves the use of a distal black rubber hood (OE-A58; Pentax) at the tip of the endoscope, to fix the distance between the tip of the endoscope and the gastric mucosa at 2 mm. The OE System will be used in mode 1 and mode 2 without optical magnification, to obtain an overview of the gastric body and identify any gross changes in the mucosa, then optical magnification will be implemented.
  Interventions: Diagnostic Test: High-definition magnification with digital chromoendoscopy.

INTERVENTIONS:
Diagnostic Test: High-Definition white light endoscopy. — evaluation of the gastric mucosa with high-definition white light endoscopy (EG-29i10 gastroscope and EPKi7010 video processor). The endoscopy images will be seen on a 27inch, flat panel, high definition LCD monitor (Radiance™ ultraSC-WU27-G1520 model) by
  Groups: High-Definition white light endoscopy.
Diagnostic Test: High-definition magnification with digital chromoendoscopy. — Subject will be evaluated by upper endoscopy with the OE System (EPK-i7010 HD Video Processor and MagniView™ EG-2990Zi Video Gastroscope) with intravenous sedation in a standardized manner. This technique involves the use of a distal black rubber hood (OE-A58; Pentax) at the tip of the endoscope, to fix the distance between the tip of the endoscope and the gastric mucosa at 2 mm. The OE System will be used in mode 1 and mode 2 without optical magnification, to obtain an overview of the gastric body and identify any gross changes in the mucosa, then optical magnification will be implemented.
  Groups: High-definition magnification with digital chromoendoscopy.

SUMMARY:
Gastric cancer is the third most common cause of cancer-related death worldwide (1). Upper endoscopy is necessary to detect neoplastic macroscopic features at an early stage, but subtle abnormalities in the gastric mucosa are often missed or misdiagnosed (1). Helicobacter pylori (Hp) is involved in the pathogenesis of gastric diseases, such as, peptic ulcers, gastric lymphoma, and gastric cancer. Therefore, the necessity to recognize malignant gastric lesions at an early stage is imperative.

DETAILED DESCRIPTION:
Previous I-SCAN™ technology uses white light as illumination light and digital post-processing of the reflection afterwards creates images yielding the virtual chromoendoscopic image. Emission of white light alone causes a potential limitation for the current I-SCAN™ technology to obtain high-quality images of microvascular patterns on the mucosal surface compared to narrow band imaging (NBI) with optical magnification.

Pentax Medical (HOYA, Tokyo, Japan) developed the Optical Enhancement™ (OE) System, which combines bandwidth-limited light with an endoscopy video system. The OE System combines digital signal processing with optical filters that limit the spectral characteristics of the illuminating light, connecting the peaks of the hemoglobin absorption spectrum (415 nm, 540 nm, and 570 nm) to create a continuous wavelength spectrum. This system has two modes that use different filters to optimize the visualization of specific features. Mode 1 is designed to improve visualization of microvessels with enough light. Mode 2 is designed to improve contrast of white-light observation by bringing the color tone of the overall image closer to that of natural color (white color tone) with more light than Mode 1 filter.

In addition, high definition optical magnification endoscopes have been developed and can combine high-definition imaging with optical magnification to produce detailed images with magnification of up to 136×. This imaging technique facilitates the evaluation of the superficial vascular aspects of the mucosa, enabling the identification of early signs of inflammation or lesions not previously seen with conventional endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* agreed to participate in the study
* patients with dyspepsia in accordance with Rome criteria

Exclusion Criteria:

* those taking NSAIDS, PPIs or antibiotics three weeks prior invitation
* severe uncontrolled coagulopathy
* prior history of gastric surgery
* those pregnant or nursing females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size was estimated with a 95% confidence interval and a 10% margin of error, based on the results of C. Robles et al. All consecutive participants will have dyspepsia according to the Rome IV criteria, and needs to be ≥18 years old. Participants need to have an epigastric pain syndrome (defined as localized pain or burning pain in the upper abdomen at least once a week, which was intermittent, nongeneralized, not relieved by defecation, and did not meet the criteria for pathology of the gallbladder or sphincter of Oddi); and/or a postprandial distress syndrome (defined as the presence of a nagging feeling of postprandial fullness after normal-volume meals, and/or early satiety that prevented the completion of a regular meal several times a week). The criteria need to be present within the 3 months prior to enrolment, and to have started ≥6 months prior to diagnosis of dyspepsia.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
1. Overall accuracy of High-definition white light endoscopy to detect lesions compatible with gastritis, H. pylori infection, gastric atrophy or intestinal metaplasia. | 3-month after index endoscopy
  histological analysis of gastritis, H. pylori infection, gastric atrophy or intestinal metaplasia.
2. Overall accuracy of optical enhancement with optical magnification to detect lesions compatible with gastritis, H. pylori infection, gastric atrophy or intestinal metaplasia. | 3-month after index endoscopy
  histological analysis of gastritis, H. pylori infection, gastric atrophy or intestinal metaplasia.
3. Comparative analysis between High-definition white light endoscopy and optical enhancement with optical magnification with histological analysis. | 1-month after finishing enrollment
  statistical analysis of the accuracy for both diagnostic methods

CONTACTS AND LOCATIONS:
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussain I, Ang TL. Evidence based review of the impact of image enhanced endoscopy in the diagnosis of gastric disorders. World J Gastrointest Endosc. 2016 Dec 16;8(20):741-755. doi: 10.4253/wjge.v8.i20.741. PMID 28042388
- [Background] Robles-Medranda C, Valero M, Puga-Tejada M, Oleas R, Baquerizo-Burgos J, Soria-Alcivar M, Alvarado-Escobar H, Pitanga-Lukashok H. High-definition optical magnification with digital chromoendoscopy detects gastric mucosal changes in dyspeptic-patients. World J Gastrointest Endosc. 2020 Jan 16;12(1):23-32. doi: 10.4253/wjge.v12.i1.23. PMID 31942231